CLINICAL TRIAL: NCT03300856
Title: Chart Review: Central Motor Conduction Time in Neurological Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999917170; 17-N-N170
Record Dates: First submitted 2017-10-03; First posted 2017-10-04 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Neurological Disorder
Keywords: Transcranial Magnetic Stimulation (TMS); Electrophysiology
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chart Review: Existing records of patients within the NINDS database who have had TMS performed to measure central motor conduction time (CMCT).

SUMMARY:
Background:

TMS stands for transcranial magnetic stimulation. It is a non-invasive way to stimulate the brain. It helps researchers study the nervous system. TMS can assess central motor conduction time (CMCT). That can be used to diagnose some diseases. It can also show how well treatments are working. Researchers want to study the records of people who have already had TMS. They want to see how it relates to the results of diagnostic studies.

Objectives:

To study the results of transcranial magnetic stimulation in certain neurological disorders. To create a descriptive analysis of the results.

Eligibility:

Records that are already in the NINDS database

Design:

The study will not enroll any participants.

Researchers will search the database for certain terms. These include TMS, CMTC, and motor evoked potentials. This will identify records of people who had TMS for diagnosis.

Using data from the records, researchers will calculate CMCT. They will note other data that relate to CMCT.

Researchers will analyze their findings. They will write a review article.

Personal data will be removed from all the records before the findings are analyzed.

DETAILED DESCRIPTION:
Objective- To retrospectively study the results of transcranial magnetic stimulation (TMS) in various neurological disorders and create a descriptive analysis of the results.

Study population- Existing records of patients within the NINDS database who have had TMS performed to measure central motor conduction time (CMCT).

Design-

* Retrospective descriptive analysis.
* The NINDS EMG Database will be queried using terms such as TMS, CMCT, and MEP (motor evoked potentials) to identify EMG reports on patients who underwent TMS for diagnosis
* Within these reports peripheral motor conduction time (PMCT), the cortical motor evoked potential (MEP) latency and amplitude will be used to calculate CMCT, clinical patient factors pertinent to estimation of CMCT as well clinically significant physical exam findings will be recorded as well.
* Clinical diagnoses and neurological exams will be extracted from medical records
* Patient identifiers will be de-linked after compiling data from medical records

Outcome measures

- Results of CMCT using TMS in different diagnoses will be summarized for different neurologic disorders and correlated to clinical exam measures documented in previous records

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patients who were seen in the NINDS EMG section for diagnostic TMS studies
  2. Patients tested between 1998 and 2017
  3. Greater than or equal to age 18.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Existing records of patients within the NINDS database who have had TMS performed to measure central motor conduction time (CMCT).
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2018-07-19 (Actual)

PRIMARY OUTCOMES:
Summary of central motor conduction studies in neurological disorders | Study completion

CONTACTS AND LOCATIONS:
Overall Officials: Mary Kay Floeter, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States